CLINICAL TRIAL: NCT05930821
Title: Exercise Training, Cognition, and Mobility in Older Adults With Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Peixuan Zheng, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-1282
Record Dates: First submitted 2023-06-07; First posted 2023-07-05 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Older Adults; Multiple Sclerosis; Cognitive Impairment; Walking Impairment
Keywords: Cognition; Walking; Exercise; Physical Activity
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction; Motor Activity | interventions — Pliability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic and Resistance Exercise Program (GEMS program) (Experimental): This intervention condition will deliver the Guidelines for Exercise in Multiple Sclerosis (GEMS) program. Participants in this condition will receive a 16-week home-based, remotely supported aerobic and resistance exercise training intervention.
  Interventions: Behavioral: Aerobic and Resistance Exercise Program (GEMS program)
- Flexibility and Stretching Program (FLEX-MS program) (Active Comparator): Participants in this condition will receive a 16-week home-based, remotely supported stretching program emphasizing flexibility and range of motion as important components of fitness based on Stretching for People with MS: An Illustrated Manual from the National MS Society.
  Interventions: Behavioral: Flexibility and Stretching Program (FLEX-MS program)

INTERVENTIONS:
Behavioral: Aerobic and Resistance Exercise Program (GEMS program) — * Remotely-coached/guided, home-based program delivered using telerehabilitation focusing on aerobic fitness and muscle strength as a mode of training.
  * The exercise training prescription involves performing 3 days per week and include (a) aerobic exercise: 30+ minutes of moderate-intensity walking (≥100 steps/min) monitored by a waist-worn pedometer, and (b) resistance training: 1-2 sets, 10-15 repetitions of 5-10 exercises targeting lower and upper body, and core muscle groups using elastic bands.
  * Other components of the GEMS program include appropriate exercise equipment (pedometer, resistance bands), one-on-one coaching sessions via Zoom, action-planning via calendars, logbooks for self-monitoring, and SCT-based newsletters.
  Arms: Aerobic and Resistance Exercise Program (GEMS program)
Behavioral: Flexibility and Stretching Program (FLEX-MS program) — * Remotely-coached/guided, home-based program delivered using telerehabilitation focusing on stretching and range of motion as the mode of training.
  * The training will involve the same frequency, duration, timeline, behavior change content, and interactions with behavioral coach as the GEMS program, and account for activity, social-contact, and attention.
  * Other components of the FLEX-MS program include appropriate exercise equipment (yoga mat), one-on-one coaching sessions via Zoom, calendars, logbooks and newsletters similar to the GEMS program.
  Arms: Flexibility and Stretching Program (FLEX-MS program)

SUMMARY:
The overall objective of the proposed randomized controlled (RCT) is to determine the feasibility and efficacy of a 16-week theory-based, remotely-delivered, combined exercise (aerobic and resistance) training intervention for improving cognitive and physical function in older adults (50+ years) with multiple sclerosis (MS) who have mild-to-moderate cognitive and walking impairment. Participants (N=50) will be randomly assigned into exercise training (combined aerobic and resistance exercise) condition or active control (flexibility and stretching) condition. The 16-week intervention will be delivered and monitored remotely within a participant's home/community and supported by Zoom-based chats guided by social cognitive theory (SCT) via a behavioral coach. Participants will receive training materials (e.g., prescriptive manual and exercise equipment), one-on-one coaching, action-planning via calendars, self-monitoring via logs, and SCT-based newsletters. It is hypothesized that the home-based exercise intervention will yield beneficial effects on cognition, mobility, physical activity, and vascular function compared with an active control condition (flexibility and stretching intervention), and these improvements will be sustained during a 16-week follow-up period.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an immune-mediated and neurodegenerative disease of the central nervous system that is markedly increasing in prevalence amongst older adults. Older adults with MS present with poor health status and functioning, cognitive and ambulatory difficulty, dependence for activities of daily living, and reduced physical activity participation. The common approach for managing MS involves disease-modifying drugs, yet this first-line approach for medical management has little efficacy in older MS age groups (i.e., those 50+ years of age). Exercise training has been recognized as a promising approach for maintaining and/or restoring physical and cognitive health in older adults from the general population and younger adults with MS. To date, there is a dearth of research examining the benefits of exercise training among older adults with MS. The current study proposes a remotely-delivered exercise training program for improving cognition and mobility among older adults with MS. The proposed research adopts an innovative intervention approach (via telerehabilitation) with rigorous design for evaluating the feasibility and efficacy of a home-based exercise intervention program in older adults with MS who have cognitive and walking impairment. This exercise training program adopts an innovative intervention approach via telerehabilitation and is convenient and accessible for older adults with MS. This research may have practical relevance for improving physical activity among older adults with MS through alleviating travel concerns and reducing environmental/social barriers. If successful, the proposed project will provide foundations for implementing larger, high-quality RCTs using remotely-delivered exercise intervention for managing the consequences of aging and MS and ultimately contributing to successful aging with MS.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older
* Diagnosis of MS
* Relapse-free for the past 30 days
* Internet and e-mail access
* Ability to travel to the laboratory (for testing only)
* Willingness to complete the assessments and be randomized
* Ambulatory with or without a single-point assistive device
* Mild-to-moderate cognitive impairment (TICS-M; MSNQ)
* Walking impairment (MSWS-12)

Exclusion Criteria:

* Individuals not meeting above inclusion criteria
* Individuals with moderate to high risk for contraindications of possible injury or death when undertaking strenuous or maximal exercise (PARQ)
* Individuals diagnosed with other neurological conditions or cardiovascular diseases

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | Changes in BICAMS test scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS); the total test scores range between 0 (min) and 236 (max), higher scores indicate better cognitive function.
Cognitive Function | Changes in NIH toolbox cognitive test scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  National Institute of Health Toolbox (NIH toolbox) with customized cognitive test battery; the scores range between 0 (min) and 186 (max), higher scores indicate better cognitive function.
Physical Function | Changes in physical function scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Short Physical Performance Battery (SPPB); the performance scores range between 0 (min) and 12 (max) points, higher scores reflect better physical function.
Lower-extremity Function | Changes in lower-extremity function scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  30-Second Sit to Stand Test (30STS). The score is the number of complete repetitions of sit-to-stand movements performed during 30 seconds; the minimum value is 0 repetitions, and the maximum value depends on individuals' performance. Higher scores reflect better lower extremity function.
Functional Mobility | Changes in functional mobility scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Timed Up and Go Test (TUG); the score is the average time (in seconds) for completing two trials. The minimum and maximum scores depend on individuals' performance; shorter time (lower scores) reflects better functional mobility.
Walking Endurance | Changes in walking endurance scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Six-Minute Walk Test (6MW); the score is the total walking distance (in meters) during the 6 minutes. The minimum value is 0 meter, and the maximum value depends on individuals' performance. A longer distance (higher scores) indicates better walking endurance.
Walking Speed | Changes in walking speed scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Timed 25-foot Walking Test (T25FW); the score is the average speed (25 feet divided by time, ft/s) for completing two trials. The minimum and maximum scores (time) depend on individuals' performance. A faster speed represents better ambulatory performance.

SECONDARY OUTCOMES:
Physical Activity Level | Changes in time spent in MVPA from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Time spent in moderate-to-vigorous physical activity (MVPA) will be measured by a waist-worn accelerometer (ActiGraph model GT3X+); a longer time (in seconds) reflects a higher level of physical activity.
Physical Activity Level | Changes in daily step count from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Daily step count will be measured by a waist-worn accelerometer (ActiGraph model GT3X+); a greater number of steps per day reflects a higher level of physical activity.
Exercise Behavior | Changes in the GLTEQ scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Godin Leisure-Time Exercise Questionnaire (GLTEQ); scores range between 0 (min) and 119 (max), higher scores indicate greater engagement in exercise behavior.
Vascular Function | Changes in central blood pressure from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Central blood pressure will be measured by waveform analysis using the SphygmoCor XCEL System. A higher value (in millimeters of mercury, or mmHg) indicate higher blood pressure.
Vascular Function | Changes in augmentation index from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Augmentation index is a biomarker for arterial stiffness and will be measured using the SphygmoCor XCEL System. A higher value (percentage) indicates greater arterial stiffness.
Vascular Function | Changes in cfPWV from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Carotid-to-femoral pulse wave velocity (cfPWV) is a biomarker for arterial stiffness and will be measured using the SphygmoCor XCEL System. A higher value (meters/second) indicates greater arterial stiffness.

OTHER OUTCOMES:
Fatigue Severity | Changes in fatigue severity scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Fatigue Severity Scale (FSS); scores range between 1 (min) and 7 (max), higher scores reflect greater fatigue severity.
Fatigue Impact | Changes in fatigue impact scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Modified Fatigue Impact Scale (MFIS); scores range between 0 (min) and 84 (max), higher scores reflect a greater impact of fatigue on daily life.
Depressive Symptoms | Changes in depressive symptoms scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.
Anxiety | Changes in anxiety scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.
Level of Pain | Changes in pain level from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Short-form McGill Pain Questionnaire (SF-MPQ); scores range between 0 (min) and 45 (max), higher scores reflect higher level of pain.
Sleep Quality | Changes in sleep quality scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Pittsburgh Sleep Quality Index (PSQI); scores range between 0 (min) and 21 (max), higher scores indicate worse sleep quality.
Health-related Quality of Life | Changes in SF-36 scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Short Form Health Status Survey (SF-36); scores range between 0 (min) and 100 (max), higher scores indicate better physical and mental aspects of quality of life.
Health-related Quality of Life | Changes in MSIS-29 scores from Baseline (pre-intervention), after 16 weeks (post-intervention), and after 32 weeks (follow-up)
  Multiple Sclerosis Impact Scale (MSIS-29); scores range between 0 (min) and 100 (max), higher scores indicate greater impact of disease on daily function (i.e. worse outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Peixuan Zheng, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng P, Phillips SA, Duffecy J, DeJonge SR, DuBose NG, Motl RW. Remotely-delivered exercise training program for improving physical and cognitive functions among older adults with multiple sclerosis: Protocol for an NIH stage-I randomized controlled trial. Contemp Clin Trials. 2024 Sep;144:107636. doi: 10.1016/j.cct.2024.107636. Epub 2024 Jul 20. PMID 39038700